CLINICAL TRIAL: NCT00857961
Title: A Phase II, Randomised, Four-way Crossover Study to Compare the Steady State Pharmacokinetics of Testosterone Following Application of Different Testosterone Metered Dose (MD) Lotion® Formulations and Doses in Hypogonadal Men
Brief Title: A Study of the Pharmacokinetics of Testosterone Metered Dose (MD)-Lotion Formulations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14271; MTE07 (Other: Acrux); I5E-MC-TSAG (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-03-04; First posted 2009-03-09 (Estimated); Results first posted 2011-01-07 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 3 mL (30 mg) of 1% Testosterone MD-Lotion (Experimental): Applied once daily for 7 days to both axilla (1.5 mL to each axilla). All study participants are randomized to each of the 4 study treatments.
  Interventions: Drug: Testosterone MD-Lotion
- 1.5 mL (30 mg) of 2% Testosterone MD-Lotion (Experimental): Applied once daily for 7 days to one axilla. All study participants are randomized to each of the 4 study treatments.
  Interventions: Drug: Testosterone MD-Lotion
- 3 mL (60 mg) of 2% Testosterone MD-Lotion (Experimental): Applied once daily for 7 days to both axilla (1.5 mL to each axilla). All study participants are randomized to each of the 4 study treatments.
  Interventions: Drug: Testosterone MD-Lotion
- 4.5 mL (90 mg) of 2% Testosterone MD-Lotion (Experimental): Applied once daily for 7 days by three doses to both axilla (2 x 1.5 mL to one axilla and 1 x 1.5 mL to the other axilla). All study participants are randomized to each of the 4 study treatments.
  Interventions: Drug: Testosterone MD-Lotion

INTERVENTIONS:
Drug: Testosterone MD-Lotion — Administered Topically
  Other Names: LY900011; Axiron

SUMMARY:
Testosterone replacement treatment is the most effective way of treating hypogonadism in men. Acrux has a propriety testosterone replacement product, Testosterone MD-Lotion and this study will evaluate pharmacokinetics of testosterone MD-Lotion formulations.The study will also assess safety of the product.

ELIGIBILITY:
Inclusion Criteria:

* Male study participants with a prior documented diagnosis of hypoandrogenism as evidenced by previously documented: Hypothalamic, pituitary or testicular disorder or a Serum testosterone less than or equal to 300 ng/dL
* Were receiving, or in the investigator's opinion were eligible to receive treatment for hypoandrogenism
* Body Mass Index (BMI) less than 35 kg/m^2
* Passed the required laboratory and physical screening tests
* Haemoglobin levels at screening greater than or equal to 13.0 g/dL
* Adequate venous access on left or right arm
* Able to communicate with study staff, understand the study information sheet and sign the written Informed Consent forms; willing to follow and comply with study procedures

Exclusion Criteria:

* Any significant history of allergy and/or sensitivity to the drug products or their excipients, including any history of sensitivity to testosterone and/or sunscreens
* Any clinically significant chronic illness or finding on screening physical exam and/or laboratory testing
* Chronic skin disorder (e.g. eczema, psoriasis) likely to interfere with transdermal drug absorption
* Men with suspected reversible hypoandrogenism (i.e. due to medications, stress)
* Any man in whom testosterone therapy is contraindicated, which included those with:

  * Known or suspected carcinoma (or history of carcinoma) of the prostate or symptoms of benign prostatic hyperplasia and/or symptoms of lower urinary obstruction,
  * Known or suspected carcinoma (or history of carcinoma) of the breast,
  * Severe liver damage i.e. cirrhosis, hepatitis or liver tumours,
  * Active deep vein thrombosis, thromboembolic disorders or a documented history of these conditions,
  * Significant cerebrovascular or coronary artery disease,
  * Known or suspected sleep apnoea,
  * Hematocrit > 51%
* Men with clinically significant prostate exam or clinically significant elevated serum prostate specific antigen (PSA) level, or age adjusted reference range of PSA values.
* Current history of drug or alcohol abuse (more than 4 standard drinks per day and/or abnormal liver function tests 3 times the upper limit of the normal range values)
* Men taking concomitant medications that affect sex hormone binding globulin (SHBG) or testosterone concentrations or metabolism, or that were cytochrome P450 inducers or inhibitors, anti-coagulants (warfarin), or diabetic medications (insulin), anti-histamines
* Men involved in sport in which there was screening for anabolic steroids
* Men with uncontrolled diabetes (hemoglobin A1c [HbA1c] greater than or equal to 10%)
* Men taking any Investigational Product, or who had received an Investigational Product within 28 days prior to screening or 5 half-lives (whichever was the longer)
* Any contraindication to blood sampling
* Study participants who planned to have a surgical procedure during the course of the study
* Study participants with a partner of child bearing potential who was not willing to use adequate contraception (i.e. condoms) for the duration of the study
* Study participants whose partners were pregnant

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-31- Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tuscon, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burbank, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Britain, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone MD-Lotion: Applied once daily for 7 days.
  All study participants received each of the 4 study treatments:
  3 mL (30 mg) of 1% Testosterone metered dose (MD)-Lotion applied to both axilla (1.5 mL to each axilla).
  1.5 mL (30 mg) of 2% Testosterone MD-Lotion applied to one axilla.
  3 mL (60 mg) of 2% Testosterone MD-Lotion applied to both axilla (1.5 mL to each axilla).
  4.5 mL (90 mg) of 2% Testosterone MD-Lotion applied by 3 doses to the axilla (2 X 1.5 mL to one axilla and 1 X 1.5 mL to the other axilla).
Period: Overall Study
Arm/Group | Testosterone MD-Lotion
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 47.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meter (kg/m^2) | 30.1 (3.2)
Average Baseline Testosterone [Mean (Standard Deviation); unit: nanograms per deciliter (ng/dL)] | 193.2 (73.9)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Total Testosterone, Dihydrotestosterone, Free Testosterone: Time of Maximal Concentration (Tmax)
Description: Tmax is the time at which the maximum concentration (Cmax) was attained during the 24 hour period on Day 7.
Time Frame: Day 7 (0, 2, 4, 8, 12, 16, 20, 24 hours) of each of the four 7 day cycles of treatment
Population: All participants received all four doses of testosterone MD-lotion.
Measure: Median (Full Range); unit: hours (h)
Groups:
- 3 mL (30 mg) of 1% Testosterone MD-Lotion; 3 mL (60 mg) of 2% Testosterone MD-Lotion: Applied once daily for 7 days to both axilla (1.5 mL to each axilla).
- 1.5 mL (30 mg) of 2% Testosterone MD-Lotion: Applied once daily for 7 days to one axilla.
- 4.5 mL (90 mg) of 2% Testosterone MD-Lotion: Applied once daily for 7 days by three doses to axilla (2 x 1.5 mL to one axilla and 1 x 1.5 mL to the other axilla).
Arm/Group | 3 mL (30 mg) of 1% Testosterone MD-Lotion | 1.5 mL (30 mg) of 2% Testosterone MD-Lotion | 3 mL (60 mg) of 2% Testosterone MD-Lotion | 4.5 mL (90 mg) of 2% Testosterone MD-Lotion
Number analyzed (Participants) | 21 | 21 | 21 | 21
hours (h)
  Total Testosterone | 8.00 [1.93 to 24.00] | 12.00 [1.95 to 23.93] | 4.25 [0.00 to 20.00] | 15.98 [1.92 to 23.97]
  Dihydrotestosterone | 8.00 [1.93 to 24.00] | 11.93 [0.00 to 23.93] | 4.25 [0.00 to 24.00] | 15.98 [0.00 to 24.00]
  Free Testosterone | 8.00 [1.93 to 24.00] | 12.00 [1.95 to 23.93] | 4.25 [0.00 to 20.00] | 15.98 [1.92 to 23.97]

2. Primary Outcome: Pharmacokinetics of Total Testosterone: Maximal Concentration (Cmax), Minimum Concentration (Cmin), and Average Concentration (Cavg)
Description: Cmax is the maximum observed serum concentration of total testosterone during the 24 hour period on Day 7. Cmin is the minimum observed serum concentration during the 24 hour period on Day 7. Cavg(0-24) is the average serum concentration calculated during the 24 hour period on Day 7. Calculated as the AUC(0-24) divided by 24 hours.
Time Frame: Day 7 (0, 2, 4, 8, 12, 16, 20, 24 hours) of each of the four 7 day cycles of treatment
Population: All participants received all four doses of testosterone-MD lotion. One study participant in the 30 mg of 2% testosterone MD-lotion was not included in any analyses dependent on testosterone/DHT concentration at 24 hours, such as AUC(0-24), Cavg, and comparison of the pre-dose with 24 hours post-dose, since a 24 hour blood sample was not collected.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | 3 mL (30 mg) of 1% Testosterone MD-Lotion | 1.5 mL (30 mg) of 2% Testosterone MD-Lotion | 3 mL (60 mg) of 2% Testosterone MD-Lotion | 4.5 mL (90 mg) of 2% Testosterone MD-Lotion
Number analyzed (Participants) | 21 | 21 | 21 | 21
ng/dL
  Cmax | 546 (266) | 430 (259) | 590 (289) | 626 (264)
  Cmin | 164 (63) | 171 (59) | 221 (101) | 238 (135)
  Cavg (n=21, n=20, n=21, n=21) | 338 (100) | 294 (150) | 389 (152) | 432 (185)

3. Primary Outcome: Pharmacokinetics of Dihydrotestosterone: Maximal Concentration (Cmax), Minimum Concentration (Cmin), and Average Concentration (Cavg)
Description: Cmax is the maximum observed serum concentration of dihydrotestosterone during the 24 hour period on Day 7. Cmin is the minimum observed serum concentration during the 24 hour period on Day 7. Cavg(0-24) is the average serum concentration calculated during the 24 hour period on Day 7. Calculated as the AUC(0-24) divided by 24 hours.
Time Frame: Day 7 (0, 2, 4, 8, 12, 16, 20, 24 hours) of each of the four 7 day cycles of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | 3 mL (30 mg) of 1% Testosterone MD-Lotion | 1.5 mL (30 mg) of 2% Testosterone MD-Lotion | 3 mL (60 mg) of 2% Testosterone MD-Lotion | 4.5 mL (90 mg) of 2% Testosterone MD-Lotion
Number analyzed (Participants) | 21 | 21 | 21 | 21
ng/dL
  Cmax | 90.7 (64.1) | 69.4 (58.6) | 96.4 (46.2) | 98.6 (46.1)
  Cmin | 33.3 (14.4) | 34.6 (26.5) | 47.8 (29.4) | 49.4 (26.7)
  Cavg (n=21, n=20, n=21, n=21) | 62.3 (34.0) | 53.0 (45.4) | 71.4 (35.1) | 76.5 (35.9)

4. Primary Outcome: Pharmacokinetics of Free Testosterone: Maximal Concentration (Cmax), Minimum Concentration (Cmin), and Average Concentration (Cavg)
Description: Cmax is the maximum observed serum concentration of free testosterone during the 24 hour period on Day 7. Cmin is the minimum observed serum concentration during the 24 hour period on Day 7. Cavg(0-24) is the average serum concentration calculated during the 24 hour period on Day 7. Calculated as the AUC(0-24) divided by 24 hours.
Time Frame: Day 7 (0, 2, 4, 8, 12, 16, 20, 24 hours) of each of the four 7 day cycles of treatment
Population: All participants received all four doses of testosterone MD-lotion. One study participant in the 30 mg of 2% testosterone MD-lotion was not included in any analyses dependent on testosterone/DHT concentration at 24 hours, such as AUC(0-24), Cavg, and comparison of the pre-dose with 24 hours post-dose, since a 24 hour blood sample was not collected.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | 3 mL (30 mg) of 1% Testosterone MD-Lotion | 1.5 mL (30 mg) of 2% Testosterone MD-Lotion | 3 mL (60 mg) of 2% Testosterone MD-Lotion | 4.5 mL (90 mg) of 2% Testosterone MD-Lotion
Number analyzed (Participants) | 21 | 21 | 21 | 21
ng/dL
  Cmax | 14.6 (7.5) | 11.3 (5.9) | 15.9 (7.8) | 16.5 (6.2)
  Cmin | 4.4 (1.7) | 4.5 (1.3) | 5.9 (2.7) | 6.4 (3.6)
  Cavg n=21, n=20, n=21, n=21) | 8.9 (2.6) | 7.6 (3.1) | 10.4 (3.9) | 11.4 (4.6)

5. Primary Outcome: Pharmacokinetics of Total Testosterone, Dihydrotestosterone, Free Testosterone: Degree of Fluctuation (DF)
Description: Degree of fluctuation in serum concentration calculated as ((Cmax-Cmin)/Cavg) x 100%.
Time Frame: Day 7 (0, 2, 4, 8, 12, 16, 20, 24 hours) of each of the four 7 day cycles of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent fluctuation in concentration
Arm/Group | 3 mL (30 mg) of 1% Testosterone MD-Lotion | 1.5 mL (30 mg) of 2% Testosterone MD-Lotion | 3 mL (60 mg) of 2% Testosterone MD-Lotion | 4.5 mL (90 mg) of 2% Testosterone MD-Lotion
Number analyzed (Participants) | 21 | 20 | 21 | 21
percent fluctuation in concentration
  Total Testosterone | 107 (55) | 84 (34) | 91 (41) | 92 (36)
  Dihydrotestosterone | 85 (47) | 68 (25) | 70 (29) | 65 (24)
  Free Testosterone | 107 (55) | 84 (34) | 91 (41) | 92 (36)

6. Primary Outcome: Pharmacokinetics of Total Testosterone, Dihydrotestosterone, Free Testosterone: Area Under the Time Concentration Curve [AUC(0-24h)]
Description: Area under the serum concentration versus time curve was calculated using the linear trapezoidal rule from time 0 to 24 hours on Day 7.
Time Frame: Day 7 (0, 2, 4, 8, 12, 16, 20, 24 hours) of each of the four 7 day cycles of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/dL
Arm/Group | 3 mL (30 mg) of 1% Testosterone MD-Lotion | 1.5 mL (30 mg) of 2% Testosterone MD-Lotion | 3 mL (60 mg) of 2% Testosterone MD-Lotion | 4.5 mL (90 mg) of 2% Testosterone MD-Lotion
Number analyzed (Participants) | 21 | 20 | 21 | 21
h*ng/dL
  Total Testosterone | 8111 (2394) | 7053 (3594) | 9332 (3639) | 10361 (4436)
  Dihydrotestosterone | 1496 (816) | 1271 (1090) | 1712 (842) | 1836 (862)
  Free Testosterone | 214 (61) | 183 (74) | 250 (94) | 275 (111)

7. Secondary Outcome: Number of Participants With Adverse Events
Description: A listing of adverse events is located in the Reported Adverse Events module.
Time Frame: Baseline through 7 days of each cycle of four treatments and follow-up (up to 38 days)
Population: All participants received all four doses of testosterone-MD lotion.
Measure: Number; unit: participants
Arm/Group | 3 mL (30 mg) of 1% Testosterone MD-Lotion | 1.5 mL (30 mg) of 2% Testosterone MD-Lotion | 3 mL (60 mg) of 2% Testosterone MD-Lotion | 4.5 mL (90 mg) of 2% Testosterone MD-Lotion
Number analyzed (Participants) | 21 | 21 | 21 | 21
participants
  Serious Adverse Events | 0 | 0 | 0 | 0
  Non-Serious Adverse Events | 4 | 5 | 6 | 5

ADVERSE EVENTS:
Arm/Group | 3 mL (30 mg) of 1% Testosterone MD-Lotion | 1.5 mL (30 mg) of 2% Testosterone MD-Lotion | 3 mL (60 mg) of 2% Testosterone MD-Lotion | 4.5 mL (90 mg) of 2% Testosterone MD-Lotion
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 4/21 | 5/21 | 6/21 | 5/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mL (30 mg) of 1% Testosterone MD-Lotion (N=21) | 1.5 mL (30 mg) of 2% Testosterone MD-Lotion (N=21) | 3 mL (60 mg) of 2% Testosterone MD-Lotion (N=21) | 4.5 mL (90 mg) of 2% Testosterone MD-Lotion (N=21)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (5) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days